CLINICAL TRIAL: NCT03725540
Title: Oropharyngeal Leak Pressure Monitoring With Baska Versus I-gel Laryngeal Mask Airway During Laparoscopic Gynecologic Surgery
Brief Title: Oropharyngeal Leak Pressure Monitoring Using Baska Versus I-gel Laryngeal Mask Airway
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hala Saad Abdel-Ghaffar, Principal Investigator, Assiut University
Other Study IDs: 17300223
Record Dates: First submitted 2018-07-28; First posted 2018-10-31 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Laryngeal Masks
Keywords: Laryngeal Masks; Oropharyngeal leak pressure; I-gel laryngeal mask airway

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- I-gel group: Patients will be anesthetized using an appropriate sized I-gel mask according to the manufacturer's recommendations after lubrication with a water-soluble lubricant.
  Interventions: Device: I-gel
- BASKA Group: Patients will be anesthetized using BASKA mask after lubrication with a water-soluble lubricant.
  Interventions: Device: Baska_mask

INTERVENTIONS:
Device: I-gel — Patients will be anesthetized using an appropriate sized I-gel mask according to the manufacturer's recommendations after lubrication with a water-soluble lubricant.
  Other Names: I-gel LMA
  Groups: I-gel group
Device: Baska_mask — Patients will be anesthetized using BASKA mask after lubrication with a water-soluble lubricant.
  Other Names: The Baska_ LMA
  Groups: BASKA Group

SUMMARY:
The use of supraglottic airway devices with a gastric emptying tube in gynecological laparoscopic surgeries is growing. In addition to their ease of placement, they have low airway morbidity along with sufficient airway pressure in the Trendelenburg position and so they have been determined as an alternative to the endotracheal tube.

DETAILED DESCRIPTION:
The Baska mask is a novel supraglottic airway device with a non-inflatable cuff, an oesophageal drainage inlet and side channels to facilitate the aspiration of gastric contents and an integrated bite-block. The Baska mask comes in four sizes, ranging from pediatric to adult. The device appeared relatively easy to insert, provided a high-quality seal with the glottic aperture and the incidence of throat discomfort appeared low.

The I-gel a single use with noninflatable cuff and drain tube is being used for airway management during anesthesia since last few years. The noninflatable cuff of I-gel is made of a soft gel-like medical grade thermoplastic elastomer. The device has a buccal cavity stabilizer, an integral bite block and an epiglottic rest with a protective ridge, which prevents down folding of epiglottis during insertion.

An oropharyngeal leak pressure or 'leak' test is commonly performed with the laryngeal mask airway to quantify the efficacy of the seal with the airway. This value is important since it indicates the feasibility of positive pressure ventilation and the degree of airway protection from supracuff soiling.

Gynecological laparoscopic surgeries are associated with a decrease in thoraco-pulmonary compliance due to pneumoperitoneum and the Trendelenburg position. Minute ventilation needs to be increased to compensate for this reduction in compliance in order to maintain end-tidal carbon dioxide during pneumoperitoneum. This increase in minute ventilation can lead to an increase in airway pressures in excess of 20 cmH2O.

ELIGIBILITY:
Inclusion Criteria:

* BMI< 30kg/m2.
* ASA physical status: I-II.
* Operation: gynecological laparoscopic surgery
* under general anesthesia of an anticipated duration<1h.

Exclusion Criteria:

* Patient refusal.
* History of cardiac disease, psychological disorders, respiratory diseases including asthma, renal or hepatic failure.
* Patients who have a high risk of regurgitation or aspiration based on a history of gastroesophageal reflux, hiatus hernia, diabetes and gross obesity.
* Neck pathology

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Females, aged 18-60 years, BMI< 30kg/m2.
  * ASA physical status: I-II.
  * Operation: gynecological laparoscopic surgery
  * under general anesthesia of an anticipated duration<1h.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Leak airway pressure | Intra-operative; after device insertion up to its removal
  cmH2O

SECONDARY OUTCOMES:
Peak airway pressure | Intra-operative; after device insertion up to its removal
  cmH2O

CONTACTS AND LOCATIONS:
Overall Officials: Hala Abdelghaffar, MD, Principal Investigator — Professor of anesthesia, faculty of medicine, Assiut university, Egypt.
Locations (1):
- woman health hospital , Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schmidbauer W, Bercker S, Volk T, Bogusch G, Mager G, Kerner T. Oesophageal seal of the novel supralaryngeal airway device I-Gel in comparison with the laryngeal mask airways Classic and ProSeal using a cadaver model. Br J Anaesth. 2009 Jan;102(1):135-9. doi: 10.1093/bja/aen319. Epub 2008 Nov 16. PMID 19011262
- [Background] Joshi NA, Baird M, Cook TM. Use of an i-gel for airway rescue. Anaesthesia. 2008 Sep;63(9):1020-1. doi: 10.1111/j.1365-2044.2008.05668.x. No abstract available. PMID 18699884
- [Background] Alexiev V, Salim A, Kevin LG, Laffey JG. An observational study of the Baska(R) mask: a novel supraglottic airway. Anaesthesia. 2012 Jun;67(6):640-5. doi: 10.1111/j.1365-2044.2012.07140.x. PMID 22563956
- [Background] Pandit JJ. If it hasn't failed, does it work? On 'the worst we can expect' from observational trial results, with reference to airway management devices. Anaesthesia. 2012 Jun;67(6):578-83. doi: 10.1111/j.1365-2044.2012.07155.x. No abstract available. PMID 22563955
- [Background] Janakiraman C, Chethan DB, Wilkes AR, Stacey MR, Goodwin N. A randomised crossover trial comparing the i-gel supraglottic airway and classic laryngeal mask airway. Anaesthesia. 2009 Jun;64(6):674-8. doi: 10.1111/j.1365-2044.2009.05898.x. PMID 19453322